CLINICAL TRIAL: NCT00229723
Title: A Phase 2 Randomised, Double-Blind, Placebo-Controlled, Multicentre Comparative Study of Gefitinib 250 mg or 500 mg (IRESSA™) Given Either Continuously or Concomitantly With Cisplatin Plus Radiotherapy for the Treatment of Patients With Previously Untreated Unresected Late Stage III/IV Non-Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: IRESSA™ (Gefitinib) With Cisplatin Plus Radiotherapy for the Treatment of Previously Untreated Unresected Late Stage III/IV Non-Metastatic Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1839IL/0706; EudraCT number 2004-000358-21; D7919C00706; NCT00099398 (obsolete NCT alias)
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-06

CONDITIONS: Neoplasms, Squamous Cell
Keywords: Head and Neck Squamous Cell Carcinoma; Head and Neck Squamous Cell Cancer; Squamous Cell Carcinoma; Squamous Cell Cancer
MeSH Terms: conditions — Neoplasms, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — Gefitinib; Cisplatin; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (7):
- 1 (Placebo Comparator): Radiation + cisplatin; followed by placebo as maintenance therapy
  Interventions: Drug: cisplatin; Radiation: radiotherapy
- 2 (Experimental): 250 mg gefitinib + radiation + cisplatin; followed by placebo as maintenance therapy
  Interventions: Drug: gefitinib (Iressa); Drug: cisplatin; Radiation: radiotherapy
- 3 (Experimental): 500 mg gefitinib + radiation + cisplatin; followed by placebo as maintenance therapy
  Interventions: Drug: cisplatin; Radiation: radiotherapy; Drug: Gefitinib (Iressa)
- 4 (Experimental): gefitinib 250 mg + cisplatin + radiotherapy; followed by gefitinib 250 mg as maintenance therapy
  Interventions: Drug: gefitinib (Iressa); Drug: cisplatin; Radiation: radiotherapy
- 5 (Experimental): gefitinib 500 mg + cisplatin + radiotherapy; followed by gefitinib 500 mg as maintenance therapy
  Interventions: Drug: cisplatin; Radiation: radiotherapy; Drug: Gefitinib (Iressa)
- 6 (Placebo Comparator): placebo + cisplatin + radiotherapy; followed by gefitinib 250 mg as maintenance therapy
  Interventions: Drug: gefitinib (Iressa); Drug: cisplatin; Radiation: radiotherapy
- 7 (Placebo Comparator): placebo + cisplatin + radiotherapy; followed by gefitinib 500 mg as maintenance therapy
  Interventions: Drug: cisplatin; Radiation: radiotherapy; Drug: Gefitinib (Iressa)

INTERVENTIONS:
Drug: gefitinib (Iressa) — 250 mg oral tablet
  Other Names: ZD1839; IRESSA
  Arms: 2; 4; 6
Drug: cisplatin — intravenous infusion
Radiation: radiotherapy — radiation therapy
Drug: Gefitinib (Iressa) — 500 mg oral tablet
  Other Names: ZD1839; Iressa
  Arms: 3; 5; 7

SUMMARY:
The primary purpose of this study is to assess the effectiveness of ZD1839 250 mg and 500 mg when given either concomitantly or as maintenance to a standard therapy of radiotherapy (X-rays) plus chemotherapy (cisplatin) in terms of local disease control (progression-free) rate at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage III or IVA squamous cell carcinoma of the head and neck
* No prior surgery or chemotherapy/biological therapy/radiation therapy
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Life expectancy of more than 12 weeks

Exclusion Criteria:

* Cancers of the nasal space, oral cavity and larynx; or certain lung diseases.
* Abnormal blood chemistry; uncontrolled respiratory, cardiac, hepatic, or renal disease; or coexisting malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2004-11; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Oncology Medical Science Director, MD, Study Director — AstraZeneca
Locations (25):
- United States (2):
  - Research Site, Aurora, Colorado
  - Research Site, Dallas, Texas
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Czechia (3):
  - Research Site, Hradec Králové
  - Research Site, Pardubice
  - Research Site, Pilsen
- Germany (4):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Münster
  - Research Site, Saarbrücken
- India (4):
  - Research Site, Bangalore
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Thiruvananthapuram
- Poland (5):
  - Research Site, Gliwice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Warsaw
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Kamenitz
- Taiwan (2):
  - Research Site, Taipei
  - Research Site, Taoynan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 226 patients from 26 centres in 8 countries were randomized to receive study medication, the first patient was enrolled into the study on 13 November 2004 and the last patient completed the study on 27 June 2008. Patients were to be followed up for a maximum of two years (± 12 weeks) after randomization.
Groups:
- Placebo/Placebo: Concomitant placebo (plus cisplatin and radiotherapy) followed by placebo as maintenance therapy
- 250mg/Placebo: Concomitant gefitinib 250 mg (plus cisplatin and radiotherapy) followed by placebo as maintenance therapy
- 500mg/Placebo: Concomitant gefitinib 500 mg (plus cisplatin and radiotherapy) followed by placebo as maintenance therapy
- 250mg/250mg: Concomitant gefitinib 250 mg (plus cisplatin and radiotherapy) followed by gefitinib 250 mg as maintenance therapy
- 500mg/500mg: Concomitant gefitinib 500 mg (plus cisplatin and radiotherapy) followed by gefitinib 500 mg as maintenance therapy
- Placebo/250mg: Concomitant placebo (plus cisplatin and radiotherapy) followed by gefitinib 250 mg as maintenance therapy
- Placebo/500mg: Concomitant placebo (plus cisplatin and radiotherapy) followed by gefitinib 500 mg as maintenance therapy
Period: Concomitant Phase
Arm/Group | Placebo/Placebo | 250mg/Placebo | 500mg/Placebo | 250mg/250mg | 500mg/500mg | Placebo/250mg | Placebo/500mg
Started | 60 (Received randomized treatment) | 24 (Received randomized treatment) | 31 (Received randomized treatment) | 31 (Received randomized treatment) | 24 (Received randomized treatment) | 34 (Received randomized treatment) | 22 (Received randomized treatment)
Completed | 50 | 19 | 25 | 26 | 22 | 31 | 19
Not Completed | 10 | 5 | 6 | 5 | 2 | 3 | 3
Not completed — Adverse Event | 4 | 2 | 5 | 2 | 0 | 1 | 2
Not completed — Objective disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical progression | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Informed consent withdrawn | 3 | 2 | 0 | 2 | 0 | 0 | 0
Not completed — Severe non-compliance | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 3 | 0 | 1 | 1 | 0 | 2 | 0
Period: Maintenance Phase
Arm/Group | Placebo/Placebo | 250mg/Placebo | 500mg/Placebo | 250mg/250mg | 500mg/500mg | Placebo/250mg | Placebo/500mg
Started | 50 | 19 | 25 | 26 | 22 | 31 | 19
Completed | 25 (Completed study on randomized treatment) | 5 (Completed study on randomized treatment) | 16 (Completed study on randomized treatment) | 9 (Completed study on randomized treatment) | 7 (Completed study on randomized treatment) | 12 (Completed study on randomized treatment) | 9 (Completed study on randomized treatment)
Not Completed | 25 | 14 | 9 | 17 | 15 | 19 | 10
Not completed — Adverse Event | 7 | 2 | 1 | 4 | 7 | 5 | 2
Not completed — Objective disease progression | 5 | 5 | 3 | 6 | 2 | 9 | 5
Not completed — Clinical progression | 4 | 1 | 2 | 2 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2 | 2 | 0 | 0 | 1
Not completed — Informed consent withdrawn | 1 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Severe non-compliance | 3 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 5 | 4 | 1 | 2 | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Placebo | 250mg/Placebo | 500mg/Placebo | 250mg/250mg | 500mg/500mg | Placebo/250mg | Placebo/500mg | Total
Number analyzed (Participants) | 60 | 24 | 31 | 31 | 24 | 34 | 22 | 226
Age Continuous [Mean (Full Range); unit: Years] | 53.1 [29 to 67] | 52.5 [21 to 73] | 53.4 [30 to 74] | 54.3 [33 to 69] | 50.8 [33 to 72] | 53.4 [45 to 70] | 54.9 [31 to 73] | 53.2 [21 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 3 | 4 | 5 | 1 | 4 | 28
  Male | 52 | 21 | 28 | 27 | 19 | 33 | 18 | 198
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian (includes Indian) | 56 | 22 | 29 | 29 | 22 | 32 | 20 | 210
  Oriental | 4 | 2 | 2 | 2 | 2 | 2 | 2 | 16
Original site of primary cancer [Number; unit: Participants]
  Oral cavity | 4 | 0 | 2 | 1 | 3 | 2 | 3 | 15
  Oropharynx | 26 | 12 | 15 | 18 | 13 | 15 | 10 | 109
  Hypopharynx | 19 | 9 | 9 | 10 | 4 | 12 | 4 | 67
  Larynx | 10 | 2 | 4 | 1 | 3 | 4 | 3 | 27
  Oropharynx / Hypopharynx | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Other | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 7
Stage of disease at entry to study [Number; unit: Participants]
  Stage III | 10 | 7 | 7 | 7 | 4 | 6 | 8 | 49
  Stage IV (All these patients had Stage IVa cancer) | 50 | 17 | 24 | 24 | 20 | 28 | 14 | 177
WHO Performance Status [Number; unit: Participants]
  0 (Normal activity) | 41 | 14 | 24 | 24 | 17 | 24 | 16 | 160
  1 (Restricted activity) | 13 | 8 | 6 | 4 | 6 | 6 | 5 | 48
  2 (in bed ≤ 50% of the time) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  3 (in bed > 50% of the time) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  4 (100% Bed ridden) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not recorded | 6 | 2 | 1 | 3 | 1 | 4 | 1 | 18

OUTCOME MEASURES:

1. Primary Outcome: Local Disease Control Rate at 2 Years
Description: A patient demonstrated local disease control at 2 years if there was no evidence of failure of treatment. Failure was defined as the patient having objective disease progression (as per RECIST) inside the original irradiated area, at an isodose level (between 20% and 95%), or death.
Time Frame: Assessed at 2 yrs. Tumour assessments (clinical & by CT/MRI) were carried out during screening & regularly throughout the study until disease progression (as defined by Response evaluation criteria in solid tumours (RECIST)).
Measure: Number; unit: Participants
Arm/Group | Placebo/Placebo | 250mg/Placebo | 500mg/Placebo | 250mg/250mg | 500mg/500mg | Placebo/250mg | Placebo/500mg
Number analyzed (Participants) | 60 | 24 | 31 | 31 | 24 | 34 | 22
Participants | 21 | 7 | 15 | 7 | 7 | 9 | 9

2. Secondary Outcome: Local Disease Control Rate at 1 Year
Description: A patient demonstrated local disease control at 1 year if there was no evidence of failure of treatment. Failure was defined as the patient having objective disease progression (as per RECIST) inside the original irradiated area, at an isodose level (between 20% and 95%), or death.
Time Frame: Assessed after 1 year. Tumour assessments (clinical and by CT/MRI) were carried out during screening & regularly throughout the study until disease progression (as defined by RECIST).
Measure: Number; unit: Participants
Arm/Group | Placebo/Placebo | 250mg/Placebo | 500mg/Placebo | 250mg/250mg | 500mg/500mg | Placebo/250mg | Placebo/500mg
Number analyzed (Participants) | 60 | 24 | 31 | 31 | 24 | 34 | 22
Participants | 27 | 8 | 16 | 13 | 10 | 14 | 10

3. Secondary Outcome: Complete Response
Description: A patient was deemed to be a complete responder if the RECIST criteria for complete response were satisfied at any time during the study.
Time Frame: Assessed at 2 years. Clinical tumour assessments and tumour assessment by CT/MRI were carried out during screening and regularly throughout the study until disease progression.
Measure: Number; unit: Participants
Arm/Group | Placebo/Placebo | 250mg/Placebo | 500mg/Placebo | 250mg/250mg | 500mg/500mg | Placebo/250mg | Placebo/500mg
Number analyzed (Participants) | 60 | 24 | 31 | 31 | 24 | 34 | 22
Participants | 28 | 7 | 11 | 13 | 6 | 14 | 11

4. Secondary Outcome: Tumour Response (Complete Response + Partial Response)
Description: A patient was deemed to be have a tumour response if the RECIST criteria for complete response or partial response were satisfied at any time during the study.
Time Frame: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo/Placebo | 250mg/Placebo | 500mg/Placebo | 250mg/250mg | 500mg/500mg | Placebo/250mg | Placebo/500mg
Number analyzed (Participants) | 60 | 24 | 31 | 31 | 24 | 34 | 22
Participants | 34 | 11 | 17 | 18 | 11 | 22 | 14

5. Secondary Outcome: Progression Free Survival
Description: Percentage of participants who are progression free at 2 years (calculated using the Kaplan-Meier method, which allows for censored observations for example those lost to follow-up). A patient is said to have progressed if they have progression of target or non-target lesions or evidence of any new lesions (as defined by RECIST).
Time Frame: Clinical tumour assessments and tumour assessment by CT/MRI were carried out during screening and regularly throughout the study until disease progression (as defined by RECIST)
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo/Placebo | 250mg/Placebo | 500mg/Placebo | 250mg/250mg | 500mg/500mg | Placebo/250mg | Placebo/500mg
Number analyzed (Participants) | 60 | 24 | 31 | 31 | 24 | 34 | 22
Percentage of participants | 41.9 | 43.1 | 58.1 | 31.2 | 43.1 | 30.0 | 42.9

6. Secondary Outcome: Overall Survival
Description: Percentage of participants who are alive at 2 years (calculated using the Kaplan-Meier method, which allows for patients who do not have complete follow-up (censored observations)).
Time Frame: Overall survival assessed at 2 years
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo/Placebo | 250mg/Placebo | 500mg/Placebo | 250mg/250mg | 500mg/500mg | Placebo/250mg | Placebo/500mg
Number analyzed (Participants) | 60 | 24 | 31 | 31 | 24 | 34 | 22
Percentage of participants | 64.6 | 60.0 | 74.8 | 43.2 | 49.4 | 48.2 | 61.1

7. Secondary Outcome: Safety and Tolerability
Time Frame: Assessed over two years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo/Placebo | 250mg/Placebo | 500mg/Placebo | 250mg/250mg | 500mg/500mg | Placebo/250mg | Placebo/500mg
Serious Adverse Events (participants affected / at risk) | 23 | 9 | 21 | 15 | 14 | 16 | 11
Other Adverse Events (participants affected / at risk) | 58 | 23 | 30 | 30 | 23 | 32 | 21
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo/Placebo | 250mg/Placebo | 500mg/Placebo | 250mg/250mg | 500mg/500mg | Placebo/250mg | Placebo/500mg
Anaemia (Blood and lymphatic system disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Febrile Neutropenia (Blood and lymphatic system disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Leukopenia (Blood and lymphatic system disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 1/24 | 1/34 | 1/22
Neutropenia (Blood and lymphatic system disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Thrombocytopenia (Blood and lymphatic system disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Cardiac Arrest (Cardiac disorders) | 3/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Cardiac Failure (Cardiac disorders) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 1/34 | 0/22
Cardiopulmonary Failure (Cardiac disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Cardio-Respiratory Arrest (Cardiac disorders) | 0/60 | 0/24 | 2/31 | 0/31 | 0/24 | 0/34 | 0/22
Myocardial Infarction (Cardiac disorders) | 1/60 | 0/24 | 1/31 | 0/31 | 1/24 | 0/34 | 1/22
Deafness Bilateral (Ear and labyrinth disorders) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Hypoacusis (Ear and labyrinth disorders) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Visual Disturbance (Eye disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Abdominal Pain Upper (Gastrointestinal disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Diarrhoea (Gastrointestinal disorders) | 0/60 | 0/24 | 3/31 | 1/31 | 0/24 | 0/34 | 0/22
Dysphagia (Gastrointestinal disorders) | 2/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Gastric Ulcer (Gastrointestinal disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Gastrointestinal Disorder (Gastrointestinal disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Haematemesis (Gastrointestinal disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Intestinal Ischaemia (Gastrointestinal disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Mouth Haemorrhage (Gastrointestinal disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Nausea (Gastrointestinal disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Oesophagitis (Gastrointestinal disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Peptic Ulcer (Gastrointestinal disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Pneumoperitoneum (Gastrointestinal disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Stomatitis (Gastrointestinal disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 1/22
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1/60 | 1/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Vomiting (Gastrointestinal disorders) | 1/60 | 1/24 | 0/31 | 1/31 | 0/24 | 0/34 | 1/22
Death (General disorders) | 2/60 | 1/24 | 0/31 | 1/31 | 2/24 | 0/34 | 0/22
Facial Pain (General disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Fatigue (General disorders) | 1/60 | 1/24 | 1/31 | 1/31 | 0/24 | 1/34 | 0/22
General Physical Health Deterioration (General disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Localised Oedema (General disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Pyrexia (General disorders) | 1/60 | 0/24 | 4/31 | 0/31 | 0/24 | 0/34 | 0/22
Sudden Death (General disorders) | 0/60 | 1/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Hepatic Failure (Hepatobiliary disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Hypersensitivity (Immune system disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Bronchitis (Infections and infestations) | 0/60 | 1/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Bronchopneumonia (Infections and infestations) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Implant Site Infection (Infections and infestations) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 1/22
Laryngitis (Infections and infestations) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 1/22
Lobar Pneumonia (Infections and infestations) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Lower Respiratory Tract Infection (Infections and infestations) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Lymph Gland Infection (Infections and infestations) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Pharyngitis (Infections and infestations) | 1/60 | 1/24 | 0/31 | 1/31 | 1/24 | 0/34 | 0/22
Pneumonia (Infections and infestations) | 4/60 | 1/24 | 1/31 | 0/31 | 1/24 | 1/34 | 1/22
Pneumonia Fungal (Infections and infestations) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Sepsis (Infections and infestations) | 0/60 | 1/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Septic Shock (Infections and infestations) | 0/60 | 1/24 | 0/31 | 0/31 | 0/24 | 0/34 | 1/22
Soft Tissue Infection (Infections and infestations) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Urinary Tract Infection (Infections and infestations) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 1/22
Fall (Injury, poisoning and procedural complications) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Femur Fracture (Injury, poisoning and procedural complications) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Radiation Mucositis (Injury, poisoning and procedural complications) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Tibia Fracture (Injury, poisoning and procedural complications) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Tracheal Obstruction (Injury, poisoning and procedural complications) | 1/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 1/22
Blood Potassium Increased (Injury, poisoning and procedural complications) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 1/22
Fibrin D Dimer Increased (Injury, poisoning and procedural complications) | 1/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Renal Function Test Abnormal (Injury, poisoning and procedural complications) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Anorexia (Metabolism and nutrition disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Cachexia (Metabolism and nutrition disorders) | 0/60 | 1/24 | 0/31 | 0/31 | 0/24 | 1/34 | 1/22
Dehydration (Metabolism and nutrition disorders) | 2/60 | 1/24 | 2/31 | 0/31 | 1/24 | 1/34 | 2/22
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0/60 | 0/24 | 1/31 | 1/31 | 1/24 | 0/34 | 0/22
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Hypoglycaemia (Metabolism and nutrition disorders) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Hypokalaemia (Metabolism and nutrition disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Hyponatraemia (Metabolism and nutrition disorders) | 2/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Neck Mass (Musculoskeletal and connective tissue disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Neck Pain (Musculoskeletal and connective tissue disorders) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Degeneration Of Uterine Fibroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Oropharyngeal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 1/22
Cerebral Artery Embolism (Nervous system disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Cerebral Haematoma (Nervous system disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Convulsion (Nervous system disorders) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Dizziness (Nervous system disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Epilepsy (Nervous system disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 1/22
Hypoxic Encephalopathy (Nervous system disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Depression (Psychiatric disorders) | 0/60 | 1/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Acute Prerenal Failure (Renal and urinary disorders) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Azotaemia (Renal and urinary disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Renal Failure (Renal and urinary disorders) | 1/60 | 0/24 | 1/31 | 1/31 | 0/24 | 0/34 | 0/22
Renal Failure Acute (Renal and urinary disorders) | 3/60 | 0/24 | 0/31 | 2/31 | 0/24 | 0/34 | 1/22
Renal Impairment (Renal and urinary disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Choking (Respiratory, thoracic and mediastinal disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/60 | 1/24 | 1/31 | 1/31 | 1/24 | 1/34 | 0/22
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1/60 | 1/24 | 1/31 | 0/31 | 0/24 | 0/34 | 0/22
Pharyngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Pharyngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 2/34 | 0/22
Stridor (Respiratory, thoracic and mediastinal disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 1/34 | 0/22
Livedo Reticularis (Skin and subcutaneous tissue disorders) | 0/60 | 1/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Rash (Skin and subcutaneous tissue disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 1/22
Aortic Thrombosis (Vascular disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Arterial Thrombosis Limb (Vascular disorders) | 0/60 | 1/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Arteriosclerosis Obliterans (Vascular disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Circulatory Collapse (Vascular disorders) | 0/60 | 0/24 | 0/31 | 1/31 | 0/24 | 0/34 | 0/22
Hypertension (Vascular disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 1/22
Hypotension (Vascular disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 0/34 | 0/22
Subclavian Artery Stenosis (Vascular disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo/Placebo | 250mg/Placebo | 500mg/Placebo | 250mg/250mg | 500mg/500mg | Placebo/250mg | Placebo/500mg
Anaemia (Blood and lymphatic system disorders) | 9/60 | 6/24 | 7/31 | 10/31 | 6/24 | 8/34 | 2/22
Leukopenia (Blood and lymphatic system disorders) | 8/60 | 5/24 | 5/31 | 6/31 | 5/24 | 7/34 | 4/22
Neutropenia (Blood and lymphatic system disorders) | 8/60 | 4/24 | 6/31 | 6/31 | 4/24 | 7/34 | 5/22
Thrombocytopenia (Blood and lymphatic system disorders) | 2/60 | 0/24 | 3/31 | 1/31 | 0/24 | 0/34 | 0/22
Atrial Fibrillation (Cardiac disorders) | 3/60 | 0/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Deafness (Ear and labyrinth disorders) | 2/60 | 0/24 | 0/31 | 1/31 | 2/24 | 0/34 | 0/22
Ear Pain (Ear and labyrinth disorders) | 6/60 | 2/24 | 0/31 | 2/31 | 0/24 | 3/34 | 0/22
Hypoacusis (Ear and labyrinth disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 1/24 | 2/34 | 0/22
Tinnitus (Ear and labyrinth disorders) | 1/60 | 0/24 | 2/31 | 1/31 | 1/24 | 1/34 | 1/22
Hypothyroidism (Endocrine disorders) | 0/60 | 0/24 | 2/31 | 0/31 | 1/24 | 0/34 | 1/22
Abdominal Pain (Gastrointestinal disorders) | 1/60 | 0/24 | 2/31 | 1/31 | 1/24 | 3/34 | 3/22
Constipation (Gastrointestinal disorders) | 16/60 | 4/24 | 8/31 | 4/31 | 4/24 | 13/34 | 9/22
Diarrhoea (Gastrointestinal disorders) | 9/60 | 4/24 | 18/31 | 10/31 | 11/24 | 4/34 | 8/22
Dry Mouth (Gastrointestinal disorders) | 25/60 | 12/24 | 14/31 | 13/31 | 12/24 | 17/34 | 16/22
Dyspepsia (Gastrointestinal disorders) | 1/60 | 0/24 | 1/31 | 1/31 | 2/24 | 0/34 | 0/22
Dysphagia (Gastrointestinal disorders) | 21/60 | 4/24 | 13/31 | 9/31 | 7/24 | 16/34 | 8/22
Gastritis (Gastrointestinal disorders) | 1/60 | 0/24 | 5/31 | 2/31 | 0/24 | 3/34 | 0/22
Glossodynia (Gastrointestinal disorders) | 0/60 | 0/24 | 0/31 | 2/31 | 0/24 | 1/34 | 1/22
Nausea (Gastrointestinal disorders) | 28/60 | 12/24 | 15/31 | 16/31 | 10/24 | 16/34 | 13/22
Odynophagia (Gastrointestinal disorders) | 3/60 | 0/24 | 4/31 | 1/31 | 3/24 | 4/34 | 2/22
Oral Discomfort (Gastrointestinal disorders) | 1/60 | 1/24 | 0/31 | 0/31 | 0/24 | 2/34 | 2/22
Oral Pain (Gastrointestinal disorders) | 6/60 | 3/24 | 4/31 | 3/31 | 1/24 | 4/34 | 0/22
Saliva Altered (Gastrointestinal disorders) | 3/60 | 0/24 | 1/31 | 0/31 | 2/24 | 0/34 | 0/22
Stomatitis (Gastrointestinal disorders) | 21/60 | 8/24 | 12/31 | 13/31 | 10/24 | 10/34 | 7/22
Vomiting (Gastrointestinal disorders) | 30/60 | 9/24 | 18/31 | 16/31 | 14/24 | 14/34 | 12/22
Asthenia (General disorders) | 4/60 | 2/24 | 1/31 | 1/31 | 2/24 | 2/34 | 1/22
Chest Pain (General disorders) | 1/60 | 1/24 | 2/31 | 2/31 | 0/24 | 1/34 | 1/22
Chills (General disorders) | 0/60 | 0/24 | 1/31 | 2/31 | 0/24 | 1/34 | 1/22
Face Oedema (General disorders) | 0/60 | 2/24 | 0/31 | 0/31 | 0/24 | 0/34 | 0/22
Fatigue (General disorders) | 7/60 | 3/24 | 8/31 | 5/31 | 2/24 | 4/34 | 3/22
Localised Oedema (General disorders) | 1/60 | 0/24 | 0/31 | 3/31 | 0/24 | 2/34 | 0/22
Oedema Peripheral (General disorders) | 2/60 | 2/24 | 2/31 | 1/31 | 1/24 | 1/34 | 0/22
Pain (General disorders) | 0/60 | 2/24 | 1/31 | 1/31 | 0/24 | 2/34 | 3/22
Pyrexia (General disorders) | 12/60 | 5/24 | 8/31 | 7/31 | 6/24 | 11/34 | 6/22
Bronchitis (Infections and infestations) | 0/60 | 2/24 | 0/0 | 0/31 | 0/24 | 0/34 | 1/22
Candidiasis (Infections and infestations) | 0/60 | 0/24 | 2/31 | 1/31 | 0/24 | 1/34 | 1/22
Cellulitis (Infections and infestations) | 0/60 | 0/24 | 0/31 | 0/31 | 2/24 | 0/34 | 0/22
Folliculitis (Infections and infestations) | 0/60 | 0/24 | 1/31 | 0/31 | 2/24 | 1/34 | 0/22
Furuncle (Infections and infestations) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 2/34 | 0/22
Implant Site Infection (Infections and infestations) | 0/60 | 0/24 | 2/31 | 1/31 | 1/24 | 1/34 | 0/22
Laryngitis (Infections and infestations) | 1/60 | 0/24 | 1/31 | 1/31 | 0/24 | 2/34 | 0/22
Lung Infection (Infections and infestations) | 0/60 | 1/24 | 0/31 | 3/31 | 1/24 | 0/34 | 0/22
Oral Candidiasis (Infections and infestations) | 2/60 | 1/24 | 1/31 | 0/31 | 2/24 | 3/34 | 0/22
Oral Fungal Infection (Infections and infestations) | 0/60 | 0/24 | 2/31 | 1/31 | 1/24 | 2/34 | 1/22
Oral Infection (Infections and infestations) | 0/60 | 0/24 | 1/31 | 0/31 | 0/24 | 2/34 | 0/22
Oropharyngitis Fungal (Infections and infestations) | 1/60 | 1/24 | 0/31 | 2/31 | 1/24 | 0/34 | 0/22
Pharyngitis (Infections and infestations) | 7/60 | 1/24 | 6/31 | 6/31 | 2/24 | 5/34 | 3/22
Rash Pustular (Infections and infestations) | 0/60 | 1/24 | 1/31 | 2/31 | 0/24 | 1/34 | 1/22
Respiratory Tract Infection (Infections and infestations) | 2/60 | 1/24 | 2/31 | 0/31 | 0/24 | 0/34 | 0/22
Rhinitis (Infections and infestations) | 1/60 | 2/24 | 2/31 | 1/31 | 1/24 | 1/34 | 1/22
Tracheostomy Infection (Infections and infestations) | 1/60 | 1/24 | 0/31 | 0/31 | 0/24 | 2/34 | 0/22
Procedural Pain (Injury, poisoning and procedural complications) | 1/60 | 2/24 | 0/31 | 3/31 | 0/24 | 2/34 | 0/22
Radiation Associated Pain (Injury, poisoning and procedural complications) | 3/60 | 1/24 | 0/31 | 4/31 | 3/24 | 2/34 | 0/22
Radiation Dysphagia (Injury, poisoning and procedural complications) | 3/60 | 4/24 | 0/31 | 3/31 | 0/24 | 3/34 | 2/22
Radiation Mucositis (Injury, poisoning and procedural complications) | 21/60 | 12/24 | 12/31 | 9/31 | 8/24 | 12/34 | 8/22
Radiation Skin Injury (Injury, poisoning and procedural complications) | 13/60 | 8/24 | 8/31 | 7/31 | 7/24 | 10/34 | 6/22
Aspartate Aminotransferase Increased (Injury, poisoning and procedural complications) | 2/60 | 0/24 | 0/31 | 2/31 | 0/24 | 0/34 | 0/22
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 1/60 | 1/24 | 2/31 | 4/31 | 1/24 | 2/34 | 1/22
Creatinine Renal Clearance Decreased (Injury, poisoning and procedural complications) | 3/60 | 0/24 | 1/31 | 2/31 | 1/24 | 0/34 | 0/22
Hepatic Enzyme Increased (Injury, poisoning and procedural complications) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 1/34 | 2/22
Weight Decreased (Injury, poisoning and procedural complications) | 13/60 | 8/24 | 9/31 | 10/31 | 9/24 | 12/34 | 7/22
Anorexia (Metabolism and nutrition disorders) | 9/60 | 2/24 | 2/31 | 7/31 | 5/24 | 4/34 | 4/22
Dehydration (Metabolism and nutrition disorders) | 4/60 | 1/24 | 4/31 | 5/31 | 1/24 | 4/34 | 2/22
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1/60 | 2/24 | 0/31 | 0/31 | 0/24 | 1/34 | 1/22
Hypercreatininaemia (Metabolism and nutrition disorders) | 0/60 | 0/24 | 2/31 | 1/31 | 1/24 | 0/34 | 0/22
Hyperuricaemia (Metabolism and nutrition disorders) | 0/60 | 0/24 | 3/31 | 0/31 | 1/24 | 0/34 | 0/22
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4/60 | 1/24 | 3/31 | 2/31 | 1/24 | 1/34 | 0/22
Hypocalcaemia (Metabolism and nutrition disorders) | 0/60 | 0/24 | 2/31 | 1/31 | 1/24 | 1/34 | 0/22
Hypokalaemia (Metabolism and nutrition disorders) | 5/60 | 4/24 | 5/31 | 2/31 | 2/24 | 2/34 | 3/22
Hypomagnesaemia (Metabolism and nutrition disorders) | 3/60 | 2/24 | 4/31 | 3/31 | 2/24 | 1/34 | 1/22
Hyponatraemia (Metabolism and nutrition disorders) | 3/60 | 0/24 | 2/31 | 3/31 | 0/24 | 2/34 | 0/22
Back Pain (Musculoskeletal and connective tissue disorders) | 0/60 | 2/24 | 2/31 | 0/31 | 0/24 | 0/34 | 2/22
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2/60 | 0/24 | 1/31 | 0/31 | 0/24 | 0/34 | 2/22
Neck Pain (Musculoskeletal and connective tissue disorders) | 1/60 | 3/24 | 1/31 | 0/31 | 0/24 | 1/34 | 2/22
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/60 | 1/24 | 0/31 | 0/31 | 3/24 | 2/34 | 2/22
Ageusia (Nervous system disorders) | 2/60 | 1/24 | 2/31 | 0/31 | 1/24 | 1/34 | 1/22
Dizziness (Nervous system disorders) | 1/60 | 2/24 | 3/31 | 2/31 | 2/24 | 3/34 | 1/22
Dysgeusia (Nervous system disorders) | 5/60 | 1/24 | 4/31 | 4/31 | 3/24 | 2/34 | 3/22
Headache (Nervous system disorders) | 4/60 | 3/24 | 2/31 | 3/31 | 2/24 | 2/34 | 1/22
Anxiety (Psychiatric disorders) | 5/60 | 3/24 | 0/31 | 2/31 | 2/24 | 2/34 | 1/22
Confusional State (Psychiatric disorders) | 0/60 | 0/24 | 2/31 | 0/31 | 1/24 | 0/34 | 0/22
Insomnia (Psychiatric disorders) | 10/60 | 4/24 | 3/31 | 4/31 | 3/24 | 2/34 | 4/22
Oliguria (Renal and urinary disorders) | 0/60 | 0/24 | 1/31 | 1/31 | 0/24 | 2/34 | 0/22
Renal Failure (Renal and urinary disorders) | 4/60 | 3/24 | 1/31 | 2/31 | 2/24 | 1/34 | 0/22
Cough (Respiratory, thoracic and mediastinal disorders) | 10/60 | 3/24 | 7/31 | 1/31 | 2/24 | 6/34 | 2/22
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5/60 | 1/24 | 3/31 | 3/31 | 4/24 | 5/34 | 3/22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6/60 | 1/24 | 2/31 | 0/31 | 1/24 | 1/34 | 1/22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/60 | 1/24 | 1/31 | 0/31 | 1/24 | 2/34 | 0/22
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 5/60 | 1/24 | 3/31 | 1/31 | 1/24 | 4/34 | 1/22
Pharyngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 10/60 | 1/24 | 6/31 | 5/31 | 1/24 | 5/34 | 5/22
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 18/60 | 3/24 | 9/31 | 7/31 | 7/24 | 7/34 | 3/22
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 6/60 | 2/24 | 3/31 | 3/31 | 3/24 | 2/34 | 1/22
Acne (Skin and subcutaneous tissue disorders) | 1/60 | 0/24 | 2/31 | 1/31 | 2/24 | 0/34 | 0/22
Alopecia (Skin and subcutaneous tissue disorders) | 6/60 | 3/24 | 3/31 | 4/31 | 3/24 | 2/34 | 4/22
Dermatitis (Skin and subcutaneous tissue disorders) | 8/60 | 4/24 | 7/31 | 4/31 | 6/24 | 6/34 | 4/22
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1/60 | 0/24 | 2/31 | 0/31 | 1/24 | 1/34 | 1/22
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0/60 | 0/24 | 0/31 | 2/31 | 0/24 | 0/34 | 0/22
Dry Skin (Skin and subcutaneous tissue disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 2/24 | 1/34 | 1/22
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0/60 | 0/24 | 0/31 | 2/31 | 0/24 | 0/34 | 0/22
Pruritus (Skin and subcutaneous tissue disorders) | 1/60 | 0/24 | 4/31 | 0/31 | 2/24 | 0/34 | 0/22
Rash (Skin and subcutaneous tissue disorders) | 3/60 | 2/24 | 11/31 | 9/31 | 2/24 | 5/34 | 5/22
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0/60 | 0/24 | 2/31 | 1/31 | 1/24 | 1/34 | 1/22
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1/60 | 2/24 | 0/31 | 0/31 | 0/24 | 1/34 | 0/22
Skin Fibrosis (Skin and subcutaneous tissue disorders) | 3/60 | 1/24 | 3/31 | 1/31 | 3/24 | 3/34 | 1/22
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3/60 | 1/24 | 2/31 | 2/31 | 2/24 | 3/34 | 1/22
Skin Reaction (Skin and subcutaneous tissue disorders) | 6/60 | 1/24 | 2/31 | 4/31 | 2/24 | 0/34 | 3/22
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0/60 | 0/24 | 0/31 | 0/31 | 0/24 | 2/34 | 0/22
Hypertension (Vascular disorders) | 5/60 | 3/24 | 1/31 | 1/31 | 1/24 | 0/34 | 2/22
Hypotension (Vascular disorders) | 2/60 | 0/24 | 2/31 | 0/31 | 0/24 | 2/34 | 0/22
Lymphoedema (Vascular disorders) | 1/60 | 0/24 | 0/31 | 0/31 | 1/24 | 2/34 | 2/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) agrees to collaborate on the contents and formation of any publication and to pay due consideration to comments and opinions offered. AstraZeneca have 30 days for final manuscript review and may require that submission for publication be delayed in order to file patent applications.